CLINICAL TRIAL: NCT01798693
Title: Nutritional Supplementation Effects on Rehabilitation Outcomes in Rotator Cuff Pathology
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Poor subject compliance and inadequate recruitment
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Abbie Smith-Ryan, PhD, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORB-12-2374
Record Dates: First submitted 2013-01-18; First posted 2013-02-26 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Rotator Cuff/Shoulder Structure and Function
Keywords: Shoulder; Supplement; Amino Acids; Collagen; Standard of Care
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (maltodextrin) (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo (maltodextrin)
- Multi-Nutrient Blend (Active Comparator): Blend of vitamins, minerals, and amino acids, given twice daily
  Interventions: Dietary Supplement: Multi-nutrient Blend

INTERVENTIONS:
Dietary Supplement: Placebo (maltodextrin)
  Arms: Placebo (maltodextrin)
Dietary Supplement: Multi-nutrient Blend
  Arms: Multi-Nutrient Blend

SUMMARY:
Rotator Injury:

* Strength/range of Motion
* ASES, VAS

DETAILED DESCRIPTION:
The addition of a nutritional therapy to a standardized physical therapy program, may expedite recovery from shoulder injury. An attractive feature of this approach is the development of an efficacious adjunct therapy that is economically superior to traditional therapy modalities and logistically feasible.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-65 years old
* Diagnosed with rotator cuff injury that will not be treated surgically

Exclusion Criteria:

* Have received a previous injection therapy (platelet-rich plasma or corticosteroid injection) within previous 6 months
* Have used the following supplements in the previous 2 weeks: Vitamin C or D, or protein supplements
* Have poorly controlled type I or type II diabetes (HgB A1C > 9.5%) or renal insufficiency (GFR < 60 ml/min).
* Have an inability to participate in rehabilitation exercises.
* Are diagnosed with arthritis, rheumatoid arthritis, or any other autoimmune or rheumatologic disease
* Have musculoskeletal pathology in a neighboring joint or structure
* Have an allergy to any component of the nutritional supplement
* Are consuming warfarin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in shoulder function, pain, strength and range of motion | Change from baseline to four, six, and twelve weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UNC Orthopedics and Exercise and Sport Medicine, Chapel Hill, North Carolina, United States